CLINICAL TRIAL: NCT00158743
Title: A Parallel, Double-blind, Placebo Controlled, Randomized Comparison of an Anti-digoxin Antibody (Digibind) Versus Placebo for the Treatment of Antepartum Patients With Severe Preeclampsia
Brief Title: Efficacy Study of Digibind for Treatment of Severe Preeclampsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BTG International Inc. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEEP
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-07

CONDITIONS: Pre-eclampsia
Keywords: Pre-eclampsia; Hypertension; Endogenous digitalis-like factor; Anti-digoxin antibody; Digibind
MeSH Terms: conditions — Pre-Eclampsia; Hypertension | interventions — Immunoglobulin Fab Fragments; digoxin antibodies Fab fragments; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Digoxin immune fab (Active Comparator): Digibind treatment plus standard of care
  Interventions: Drug: Anti-digoxin antibody (FAB fragment)
- placebo (sodium chloride) (Placebo Comparator)
  Interventions: Other: sodium chloride

INTERVENTIONS:
Drug: Anti-digoxin antibody (FAB fragment) — intravenous administered, dose based on weight (assuming 4ng/mL EDLF concentration). Dose every 6 hours x 48 hours.
  Other Names: Digibind
  Arms: Digoxin immune fab
Other: sodium chloride
  Arms: placebo (sodium chloride)

SUMMARY:
The purpose of this study is to determine whether a commercially available anti-digoxin antibody, Digibind, can delay delivery in patients with severe pre-eclampsia. If so, this would allow more time for maternally administered steroids to prevent the development of respiratory complications in premature infants.

DETAILED DESCRIPTION:
Preeclampsia (PE) is a serious complication of third trimester pregnancy manifested by high blood pressure, proteinuria, edema, encephalopathy sometimes with seizures, and hepatic failure. There is no known specific treatment, although palliative measures such as antihypertensive drugs, magnesium, steroids and early delivery improve outcomes. Multiple abnormalities have been demonstrated in PE but the relation of these abnormalities to the cause, pathophysiology and treatment is unknown. One of these abnormalities is elevation in the circulating level of a "digoxin-like" factor (EDLF), an unknown substance that cross reacts with digoxin antibodies and inhibits Na,K ATPase. An extensive literature supports the hypothesis that increased levels of EDLF may be a causative factor in the pathogenesis of hypertension. Increased levels of this factor are found both in maternal and fetal blood, both in normal pregnancy, and in pregnancy complicated by PE. Levels of this factor are higher in PE than in normal pregnancy suggesting it might play a role in the pathophysiology of PE.

Digibind (Glaxo Smith Kline) is a commercially available FAB fragment, antidigoxin antibody approved for the treatment of digoxin intoxication. In experimental models of hypertension with elevated EDLF levels, Digibind has been shown to lower blood pressure, suggesting that the antibody cross reacts with EDLF. These observations have led to the hypothesis that Digibind might ameliorate some of the manifestations of PE, especially the hypertension. Based on an extensive pre-clinical literature supporting that hypothesis, and encouraging results in 8 cases, a clinical trial is planned to test the effect of Digibind in severe PE. The study is a multi- site, parallel, double blind, placebo controlled, randomized trial. After randomization, 50 patients will be given the usual treatment for severe PE, plus study drug (Digibind or placebo) every six hours, for 48 hours. The study may be terminated during the treatment period for standard indications for early delivery.

Data collection will include: delivery latency, maternal blood pressure, antihypertensive use, renal function, hepatic function, CBC and platelet count, and umbilical artery blood flow by color doppler. Standard maternal and fetal monitoring will be followed. Newborn assessment will include: status at birth, APGAR score, NICU length of stay, respirator use and duration, and any medical complications. Adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* A subject with a diagnosis of severe preeclampsia will be eligible for inclusion if she meets the following criteria:

  1. In the opinion of the investigator delivery is considered to be probably required within a 72 hour time period and, therefore, corticosteroid administration is needed.
  2. Meets both American College of Obstetricians (ACOG) criteria for preeclampsia (modified to limit selection to patients with the required severity)

     * A systolic blood pressure of 140 mm Hg or higher or a diastolic blood pressure of 90 mm Hg or higher occurring after 20 weeks of gestation in a woman whose blood pressure has previously been normal;
     * Proteinuria, with excretion of 0.3 g or more of protein in a 24-hour urine specimen or a urine dipstick reading of 1+ or more.
  3. Meets at least one of the following ACOG criteria for severe preeclampsia (modified to limit selection to patients with the required severity)

     . Proteinuria of 5 grams or higher in a 24-hour specimen or 3+ or greater on 2 random urine samples collected at least 4 hours apart
     * A systolic blood pressure of 160 mm Hg or higher or a diastolic blood pressure of 110 mm Hg or higher on two occasions six or more hours apart in a pregnant woman who is on bed rest;
     * Oliguria, with excretion of less than 500 ml of urine in 24 hours or average of ≤ 25 ml/hour over a 3 hour period;
     * Pulmonary edema;
     * Impairment of liver function [AST(SGOT) > 72 U/L or ALT(SGPT) > 72 U/L or LDH > 600 U/L or Total Bilirubin >1.2 mg/DL)];
     * Visual or cerebral disturbances;
     * Decreased platelet count (≥50,000/mm3 and ≤ 100,000/mm3).
  4. Has a fetal gestational age of 23 5/7 to 34 weeks.

Exclusion Criteria:

1. Is in need of immediate delivery as soon as clinically appropriate
2. Eclampsia
3. Significant antecedent obstetrical problems which may interfere with study assessments or safe participation in the study
4. Evidence of non-reassuring fetal well being
5. Evidence of lethal fetal anomaly
6. Antecedent hypertension (hypertension secondary to preeclampsia, treated or untreated is allowed)
7. Antecedent renal, hepatic, or autoimmune disease
8. Medical or psychiatric disorder which is unstable or which might interfere with study assessments or safe participation in the study
9. Evidence on medical history/evaluation of use of or need for digitalis-like products currently or in the future
10. History of a severe allergic reaction to previous medication, severe asthma, or atopy. (Patients with a history of allergic reactions to antibiotics, papain, chymopapain, or other papaya extracts may be more susceptible to allergic reactions to Digibind®)
11. Prior use of antibodies/FAB fragments from sheep (e.g. Digibind®, DigiFab, CroFab)
12. Serum creatinine ≥ 1.5 mg/dl
13. Platelet count <50,000/mm3
14. Patient intends to breast feed and does not agree to wait for a minimum of seven days after the last Digibind® dose (a breast pump would be used for this seven day period)
15. Inability to understand and provide informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vardaman M Buckalew, MD, Study Chair — Wake Forest University Health Sciences
Locations (8):
- United States (8):
  - University of South Alabama, Mobile, Alabama
  - Phoenix Perinatal Associates, Phoenix, Arizona
  - Winnie Palmer Hospital, Orlando, Florida
  - Department of Obstetrics and Gynecology, Louisiana State University Health Sciences Center, PO Box 33932, 1501 Kings Highway, Shreveport, Louisiana
  - St Mary's Health Center, St Louis, Missouri
  - Medical University of South Carolina, 96 Jonathan Lucas Street, Suite 634, PO Box 250619, Charleston, South Carolina
  - Department of OB-GYN, Division of Maternal Fetal Medicine, University of Texas Medical Branch, 301 University Boulevard, Galveston, Texas
  - St Mark's Hospital, Salt Lake City, Utah

REFERENCES:
- [Background] Adair CD, Buckalew V, Taylor K, Ernest JM, Frye AH, Evans C, Veille JC. Elevated endoxin-like factor complicating a multifetal second trimester pregnancy: treatment with digoxin-binding immunoglobulin. Am J Nephrol. 1996;16(6):529-31. doi: 10.1159/000169054. PMID 8955766
- [Background] Gusdon JP Jr, Buckalew VM Jr, Hennessy JF. A digoxin-like immunoreactive substance in preeclampsia. Am J Obstet Gynecol. 1984 Sep 1;150(1):83-5. doi: 10.1016/s0002-9378(84)80114-3. PMID 6540989
- [Background] Poston L, Morris JF, Wolfe CD, Hilton PJ. Serum digoxin-like substances in pregnancy-induced hypertension. Clin Sci (Lond). 1989 Aug;77(2):189-94. doi: 10.1042/cs0770189. PMID 2548800
- [Background] Graves SW, Williams GH. An endogenous ouabain-like factor associated with hypertensive pregnant women. J Clin Endocrinol Metab. 1984 Dec;59(6):1070-4. doi: 10.1210/jcem-59-6-1070. PMID 6092405
- [Background] Lopatin DA, Ailamazian EK, Dmitrieva RI, Shpen VM, Fedorova OV, Doris PA, Bagrov AY. Circulating bufodienolide and cardenolide sodium pump inhibitors in preeclampsia. J Hypertens. 1999 Aug;17(8):1179-87. doi: 10.1097/00004872-199917080-00018. PMID 10466474
- [Background] Krep H, Price DA, Soszynski P, Tao QF, Graves SW, Hollenberg NK. Volume sensitive hypertension and the digoxin-like factor. Reversal by a Fab directed against digoxin in DOCA-salt hypertensive rats. Am J Hypertens. 1995 Sep;8(9):921-7. doi: 10.1016/0895-7061(95)00181-N. PMID 8541008
- [Background] Krep HH, Graves SW, Price DA, Lazarus M, Ensign A, Soszynski PA, Hollenberg NK. Reversal of sodium pump inhibitor induced vascular smooth muscle contraction with digibind. Stoichiometry and its implications. Am J Hypertens. 1996 Jan;9(1):39-46. doi: 10.1016/0895-7061(95)00260-x. PMID 8834705
- [Background] Gruber KA, Whitaker JM, Buckalew VM Jr. Endogenous digitalis-like substance in plasma of volume-expanded dogs. Nature. 1980 Oct 23;287(5784):743-5. doi: 10.1038/287743a0. No abstract available. PMID 6253813

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: sodium chloride placebo
Period: Overall Study
Arm/Group | Digoxin Immune Fab | Placebo
Started | 24 | 27
Completed | 15 | 20
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Digoxin Immune Fab | Placebo | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (7.1) | 26 (6.2) | 26 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 12 | 19
  White | 10 | 7 | 17
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Creatinine Clearance
Description: change from baseline in creatinine clearance measured at 24 to 48 hours, comparing patients who received placebo with those who received digoxin immune fab
Time Frame: Baseline to 24-48 hours.
Measure: Mean (Standard Deviation); unit: milliliters/minute
Arm/Group | Digoxin Immune Fab | Placebo
Number analyzed (Participants) | 15 | 20
milliliters/minute | -8 (43) | -22 (56)

ADVERSE EVENTS:
Arm/Group | Digoxin Immune Fab | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/27
Other Adverse Events (participants affected / at risk) | 1/24 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digoxin Immune Fab (N=24) | Placebo (N=27)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digoxin Immune Fab (N=24) | Placebo (N=27)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
hypothermia (General disorders) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
uterine atony (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No